CLINICAL TRIAL: NCT06401772
Title: The Effectiveness and Safety of Body Posture to Improve Intracranial Pressure in Preventing Postoperative Recurrence for Chronic Subdural Hematoma (BP-CSDH) -A Multicenter Randomized Controlled Clinical Trial
Brief Title: The Effectiveness and Safety of Body Posture in Preventing Postoperative Recurrence for Chronic Subdural Hematoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xuehai Wu, Professor, Huashan Hospital, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2024-599
Record Dates: First submitted 2024-04-27; First posted 2024-05-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Chronic Subdural Hematoma; Recurrence
Keywords: Chronic Subdural Hematoma; body posture; intracranial pressure
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence | interventions — Posture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- body posture group (Experimental): During post-operative hospitalization, patients will receive routine treatment and keep Intracranial Hypotension Targeted (IHT) Body Posture as long as possible, with the maximum to 14 to 18 hours daily.Body Posture education for patients after discharge, which is keeping IHT Body Posture when on bed rest and sleeping within 3 months as long as possible and recording time every day.Specifically, IHT therapy requires CSDH patients to raise their lower limbs 30° higher over the horizontal level of their head. All leg-lift pads were customized from the same manufacturer and provided to participants by the research group. For patients with unilateral CSDH, the head should be tilted towards the hematoma affected side and opposite side lying should be avoided as much as possible. For patients with bilateral CSDH, there is no need for the head lateralization. To avoid food reflux and aspiration pneumonia, IHT therapy was strictly prohibited within 2 hours after each meal.
  Interventions: Behavioral: Intracranial Hypotension Targeted(IHT) Body Posture
- control group (No Intervention): Patients will be required to keep supine position. In addition to IHT Body Posture, patients will receive treatment as same as body posture group.

INTERVENTIONS:
Behavioral: Intracranial Hypotension Targeted(IHT) Body Posture — IHT therapy requires CSDH patients to raise their lower limbs 30° higher over the horizontal level of their head.For patients with unilateral CSDH, the head should be tilted towards the hematoma affected side and opposite side lying should be avoided as much as possible. For patients with bilateral CSDH, there is no need for the head lateralization.To avoid food reflux and aspiration pneumonia, IHT therapy was strictly prohibited within 2 hours after each meal
  Arms: body posture group

SUMMARY:
This study aims to investigate the effectiveness and safety of body posture to improve intracranial pressure in preventing postoperative recurrence for chronic subdural hematoma

DETAILED DESCRIPTION:
This study is a multicenter prospective randomized clinical trial with open-label treatment and blinded outcome assessment to evaluate the effects of body posture on hematoma recurrence. Patients will be assigned in a 1:1 ratio to body posture group(upper body lay flat, lower body elevate 30° or 20-30cm, head turn to affected side) or control group(supine position) randomly. After operation, patients will be required to keep respective body posture at sleep time for 3 months. Instead of body posture, patients will receive routine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. chronic hematoma is diagnosed with CT/MRI scan; thickness of hematoma is more than 1 cm;
2. more than 60 years of age or 60 years;
3. MGS-GCS (Markwalder's Grading Scale and Glasgow Coma Scale) is less than or equal to 2;
4. patients have neurological symptom caused by CSDH before surgery, such as headache, dizziness, nausea, vomiting, numbness or weakness of limb, instability to walk, unconsciousness, trouble speaking, insensitive, etc.
5. receive burr hole drainage;
6. sign informed consent voluntarily.

Exclusion Criteria:

1. pregnancy or lactation;
2. have hernia of brain or acute massive cerebral infarction that have to perform craniotomy
3. have serous cancer, hemorrhagic disease, cardiac dysfunction and other serious disease that may aggravate patient's condition and impact follow-up;
4. patients can not stay in bed for long-term due to mental illness or spinal disease(kyphotic deformity);
5. CT scan showed that no obvious brain compression or midline shift; no symptom before surgery; neurosurgeon evaluate that patients do not require surgery;
6. have CSDH for more than 1 year or organized hematoma;
7. CSDH caused by over V-P shunting;
8. during burr hole drainage, patients have to perform craniotomy due to acute bleeding or brain hernia;
9. during burr hole drainage, patients have cerebral contusion or drainage catheter insert into brain unexpectedly;
10. have venous thrombosis of lower extremity or pulmonary embolism;
11. cannot regular reexamine within 1 year for any reason;
12. life expectancy less than 1 year;
13. participating other ongoing clinical trial;
14. patients are not qualified for other reason evaluated by two neurosurgeons;
15. have bile reflux gastritis and esophageal diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
subdural hematoma recurrence rate | within 90±10 days post-surgery
  Recurrence is defined as maximum thickness of subdural hematoma more than 10mm, and patients have subdural hematoma related symptoms without head injury.

SECONDARY OUTCOMES:
change in modified Rankin Scale(mRS) compared to baseline | 90days and 1year post-surgery
  The mRS is a clinician-reported measure of global disability,ranging from 0 to 6, with higher scores indicating more severe disability
change in EQ-5D-5L score compared to baseline | 90days and 1year post-surgery
  The 5-level EQ-5D version (EQ-5D-5L) is a standardised measure of health status
differences between two group in comorbidities | 90days post-surgery
  comparison of comorbidities rate of two group
differences between two group in complications | 90day post-surgery
  comparison of complications rate of two group
subdural hematoma recurrence rate | 1year post-surgery
  comparison of recurrence rate of two group
all cause recurrence rate | 90days and 1year post-surgery
  comparison of recurrence rate of two group caused by whatever the reasons
differences between two group in recurrence time | within 90days and 1year post-surgery
  comparison of recurrence time of two group

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Wu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University; ying mao, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No